CLINICAL TRIAL: NCT02886078
Title: Dorsal Versus Volar Approach for CapFlex-PIP© Implantation: a Randomized Controlled Trial
Brief Title: Dorsal Versus Volar Approach for CapFlex-PIP© Implantation
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Insufficient recruitment
Sponsor: Miriam Marks (Other)
Responsible Party: Sponsor-Investigator, Miriam Marks, Dr. phil., Schulthess Klinik
Organization: Schulthess Klinik (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CapFlexRCT
Record Dates: First submitted 2016-08-23; First posted 2016-09-01 (Estimated); Last update posted 2017-06-16 (Actual); Status verified 2017-06

CONDITIONS: Osteoarthritis
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dorsal approach CapFlex arthroplasty (Experimental): Arthroplasty of the PIP joint with the CapFlex implant. Surgery will be done with the dorsal approach.
  Interventions: Procedure: Dorsal approach CapFlex arthroplasty
- Volar approach CapFlex arthroplasty (Active Comparator): Arthroplasty of the PIP joint with the CapFlex implant. Surgery will be done with the volar approach.
  Interventions: Procedure: Volar approach CapFlex arthroplasty

INTERVENTIONS:
Procedure: Dorsal approach CapFlex arthroplasty — Arthroplasty of the PIP joint with the CapFlex implant. Surgery will be done with the dorsal approach.
  Arms: Dorsal approach CapFlex arthroplasty
Procedure: Volar approach CapFlex arthroplasty — Arthroplasty of the PIP joint with the CapFlex implant. Surgery will be done with the volar approach.
  Arms: Volar approach CapFlex arthroplasty

SUMMARY:
The primary objective is to investigate the active extension six months after implantation of the CapFlex-PIP© arthroplasty, comparing the dorsal with the volar approach.

This is a randomized controlled trial including 70 patients with PIP OA indicated for CapFlex arthroplasty.

DETAILED DESCRIPTION:
The CapFlex-PIP© implant is a modular gliding surface proximal interphalangeal (PIP) joint prosthesis. For implantation, there are two approaches available: The dorsal central split approach according to Swanson and the volar approach described by Simmen.

Our experiences and data from our prospective registry indicate, that the active extension of the PIP joint is better after the dorsal approach, but sometimes related with hyperextension of the PIP joint and secondary swan-neck deformity. Extension is supposed to be better after the volar approach, but associated with active and passive extension lag. Evidence of theses experiences will assist the surgeon in the preoperative planning to select the appropriate approach according to the patient's needs.

The primary objective is to investigate the active extension six months after implantation of the CapFlex-PIP© arthroplasty, comparing the dorsal with the volar approach.

This is a randomized controlled trial.

ELIGIBILITY:
Inclusion Criteria:

* Indication for CapFlex-PIP© arthroplasty
* Patient aged 18 years and over
* Informed Consent as documented by signature

Exclusion Criteria:

* Revision surgery
* CapFlex-PIP© arthroplasty at the thumb IP joint
* Major surgery at the same finger (e.g. DIP arthrodesis)
* Ulnar/radial deviation of the PIP joint > 15°
* Patients in which a reconstruction of the collateral ligaments has to be performed
* General medical contraindication to surgery
* German language barrier to complete the questionnaires
* Any disease process that would preclude accurate evaluation (e.g. neuromuscular, psychiatric or metabolic disorder)
* Pregnancy
* Surgery not planned by Dr. Herren, Dr. Schindele or Dr. Bodmer
* Legal incompetence

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Active extension of the PIP joint measured with a goniometer | 6 months after surgery

SECONDARY OUTCOMES:
Subjective function using the Brief Michigan Hand Questionnaire (briefMHQ) | 6 months after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Schulthess Klinik, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No
No plan to share data